CLINICAL TRIAL: NCT05990335
Title: Mobile Software Application Intervention Including Cognitive Tasks
Brief Title: Boost Study 21270 (Cognition)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NXTech (Industry)
Collaborators: Kansas State University (Other); National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: NX-21270; R43DA051270 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Function Abnormal
Keywords: Cognition
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: Between subjects and within subjects mixed design, reflecting major variables of high/low group intervention/control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognition exercises group I (Experimental): Subjects enrolled in this arm are exposed to an active task intervention designed for higher cognitive effort training functions
  Interventions: Behavioral: mHealth application (custom)
- Cognition exercises group C (Active Comparator): Subjects enrolled in this arm are exposed to an active task intervention designed for lower cognitive effort training functions
  Interventions: Behavioral: mHealth application (custom)

INTERVENTIONS:
Behavioral: mHealth application (custom) — Smartphone based application designed to engage user executive functions

SUMMARY:
This study is designed to to test the technical feasibility of encouraging interaction with a mobile smartphone software package (mHealth app) for training aspects of executive function and cognition.

DETAILED DESCRIPTION:
The purpose of this human subjects study is to test the technical feasibility of interaction with a mobile smartphone software package (mHealth app) for training in aspects of executive function and cognition. The study participants are healthy subjects recruited online, with consent secured at the time of screening, and with enrollees assigned to High or Low groups on the basis of initial screening task scores. Subjects are requested to participate in directed interaction activities for up to 8 weeks, with measures primarily evaluating feasibility of MHealth app package task completion and secondarily evaluating the cognitive effect of activities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Fluent in English
* Resides in the United States
* Score on prescreen task is in 25% quartile
* Familiar with smartphone device app installation and device usage
* Possesses a compatible smartphone

Exclusion Criteria:

None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Smith, Study Director — Kansas State
Locations (1):
- Kansas State DPS, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognition Exercises Group I | Cognition Exercises Group C
Started | 64 | 60
Completed | 64 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Units are participants are population is same as assignment in Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognition Exercises Group I | Cognition Exercises Group C | Total
Number analyzed (Participants) | 64 | 60 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 60 | 123
  >=65 years | 1 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 17 | 26 | 43
  Female | 37 | 29 | 66
  Transgender Male or Transgender Female | 3 | 1 | 4
  Not Reported | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 7 | 8
  Black / African American | 6 | 4 | 10
  Hispanic | 6 | 9 | 15
  White | 41 | 36 | 77
  Unreported | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64 | 60 | 124

OUTCOME MEASURES:

1. Primary Outcome: Task Completion Rate
Description: Percentage of participants completing minimum required weekly interactions
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: Percentage of eligible participants
Arm/Group | Cognition Exercises Group I | Cognition Exercises Group C
Number analyzed (Participants) | 64 | 60
Percentage of eligible participants | 66 (15) | 57 (19)

2. Secondary Outcome: Change in Task Performance
Description: Change in Human Hypothetical Choice scale (higher scores indicate a better outcome, minimum value 0 to maximum value 1), calculated as value at 8 weeks minus value at 1 week
Time Frame: At 8 weeks
Population: Subgroup of participants in each arm completing all study weeks and requested activities, were analyzed
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognition Exercises Group I | Cognition Exercises Group C
Number analyzed (Participants) | 21 | 29
units on a scale | 0.62 (0.03) | 0.62 (0.04)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Cognition Exercises Group I | Cognition Exercises Group C
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/60
Other Adverse Events (participants affected / at risk) | 0/64 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT05990335/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT05990335/SAP_001.pdf